CLINICAL TRIAL: NCT01381887
Title: A Double-Blind, Placebo-Controlled, Randomized, Crossover, Multicenter Study to Evaluate the Effect of JNJ-28431754 (Canagliflozin) on Post-Meal Glucose in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of JNJ-28431754 (Canagliflozin) on Post-Meal Glucose in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR018373; 28431754DIA1045
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Placebo; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Placebo Comparator): Placebo Treatment A: Form=capsule route=oral administration. Capsule is taken once daily on Day 1 and Day 2 in 1 of 4 treatment periods.
  Interventions: Drug: Placebo
- 002 (Experimental): Canagliflozin 300mg/Placebo Treatment B: Type=1 unit=mg number=300 form=capsule route=oral use. Capsule is taken once on Day 1 in 1 of 4 treatment periods.
  Form=capsule route=oral administration. Capsule is taken once on Day 2 in 1 of 4 treatment periods.
  Interventions: Drug: Canagliflozin 300mg/Placebo
- 003 (Experimental): Canagliflozin 300mg Treatment C: Type=1 unit=mg number=300 form=capsule route=oral use. Capsule is taken once daily on Day 1 and Day 2 in 1 of 4 treatment periods.
  Interventions: Drug: Canagliflozin 300mg
- 004 (Experimental): Canagliflozin 300mg/Canagliflozin 150mg Treatment D: Type=1 unit=mg number=300 form=capsule route=oral use. Capsule is taken once on Day 1 in 1 of 4 treatment periods.
  Type=1 unit=mg number=150 form=capsule route=oral use. Capsule is taken once on Day 2 in 1 of 4 treatment periods.
  Interventions: Drug: Canagliflozin 300mg/Canagliflozin 150mg

INTERVENTIONS:
Drug: Placebo — Treatment A: Form=capsule, route=oral administration. Capsule is taken once daily on Day 1 and Day 2 in 1 of 4 treatment periods.
  Arms: 001
Drug: Canagliflozin 300mg/Placebo — Treatment B: Type=1, unit=mg, number=300, form=capsule, route=oral use. Capsule is taken once on Day 1 in 1 of 4 treatment periods.
  Form=capsule, route=oral administration. Capsule is taken once on Day 2 in 1 of 4 treatment periods.
  Arms: 002
Drug: Canagliflozin 300mg/Canagliflozin 150mg — Treatment D: Type=1, unit=mg, number=300, form=capsule, route=oral use. Capsule is taken once on Day 1 in 1 of 4 treatment periods.
  Type=1, unit=mg, number=150, form=capsule, route=oral use. Capsule is taken once on Day 2 in 1 of 4 treatment periods.
  Arms: 004
Drug: Canagliflozin 300mg — Treatment C: Type=1, unit=mg, number=300, form=capsule, route=oral use. Capsule is taken once daily on Day 1 and Day 2 in 1 of 4 treatment periods.
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the effect of canagliflozin on post-meal glucose blood levels in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This is a double-blind (neither study staff or the patient will know the identity of the treatment assigned) study of canagliflozin in patients with Type 2 Diabetes Mellitus (T2DM) who are currently taking metformin at a stable dose of >=1500 mg/day. Patients will participate in the study for up to approximately 16 weeks. During the study, patients will receive 4 treatments (A, B, C, and D); each treatment will be administered during a 3-day treatment period. Patients will receive 1 dose of study medication in the morning of Day 1 and Day 2 of each treatment period and treatment periods will be separated by approximately 2 weeks. Treatments will consist of placebo (A), canagliflozin 300 mg and placebo (B), canagliflozin 300mg (C), and canagliflozin 300mg and canagliflozin 150mg (D).

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM with inadequate glycemic control (based upon fasting glucose measurements >=130 mg/dL and <=250 mg/dL) on metformin monotherapy or on metformin in dual combination with other glucose lowering agents (sulphonylurea [SU] or a meglitinide or a dipeptidyl peptidase-4 [DPP-4] inhibitor) are eligible for enrollment in the study.

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* history of a severe hypoglycemic episode within 6 months before screening
* Has repeated (ie, 2 or more over a 1-week period) fasting plasma glucose (FPG) and/or fasting self-monitored blood glucose (SMBG) measurements >=250 mg/dL (13.88 mmol/L) during the pre-treatment phase, despite reinforcement of diet and exercise counseling
* History of or current illness considered to be clinically significant by the investigator

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of glucose | Up to Day 44

SECONDARY OUTCOMES:
Rate of insulin secretion | Up to Day 44
Urinary glucose excretion (UGE) | Up to Day 44
Renal threshold of glucose excretion (RTG) | Up to Day 44
Adverse events | Up to approximately Day 44

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (5):
- United States (5):
  - Chula Vista, California
  - Miramar, Florida
  - Cincinnati, Ohio
  - Dallas, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Stein P, Berg JK, Morrow L, Polidori D, Artis E, Rusch S, Vaccaro N, Devineni D. Canagliflozin, a sodium glucose co-transporter 2 inhibitor, reduces post-meal glucose excursion in patients with type 2 diabetes by a non-renal mechanism: results of a randomized trial. Metabolism. 2014 Oct;63(10):1296-303. doi: 10.1016/j.metabol.2014.07.003. Epub 2014 Jul 9. PMID 25110280
- See also: A Double-Blind, Placebo-Controlled, Randomized, Crossover, Multicenter Study to Evaluate the Effect of JNJ-28431754 (canagliflozin) on Post-Meal Glucose in Subjects With Type 2 Diabetes Mellitus — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1114&filename=CR018373_CSR.pdf